CLINICAL TRIAL: NCT05217069
Title: Avelumab Added to FOLFIRI Plus Cetuximab Followed by Avelumab Maintenance in Patients With Previously Untreated RAS Wild-type Colorectal Cancer. The Phase II FIRE-6 Study
Brief Title: FOLFIRI + Cetuximab + Avelumab RAS Wild-type CRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); ClinAssess GmbH (Industry)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Director CCC-Munich, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIRE-6
Record Dates: First submitted 2019-01-22; First posted 2022-02-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Treatment Related Cancer
Keywords: CRC; Avelumab; FIRE; RAS
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — Fluorouracil; Leucovorin; Irinotecan; Cetuximab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RAS wild-type Avelumab (Other): Induction therapy:
  FOLFIRI 5-FU: 400 mg/m2 (i.v. bolus) Folinic acid: 400mg/m2 Irinotecan: 180 mg/m2 5-FU: 2.400 mg/m2 (i.v. 46h)
  Cetuximab 400 mg/m2 i.v. 120min initial dose 250 mg/m2 i.v. 60min q 1w
  Maintenance therapy:
  Avelumab 10mg/kg IV (day 1 q2w)
  Interventions: Drug: 5-FU; Drug: Folinic Acid; Drug: Irinotecan; Drug: Cetuximab; Drug: Avelumab

INTERVENTIONS:
Drug: 5-FU — 400 mg/m2 (i.v. bolus) 2400 mg/m2 (i.v. 46h)
Drug: Folinic Acid — 400mg/m2
Drug: Irinotecan — 180 mg/m2
Drug: Cetuximab — 400 mg/m2 i.v. 120min initial dose 250 mg/m2 i.v. 60min q 1w
Drug: Avelumab — 10mg/kg IV (day 1 q2w)

SUMMARY:
Within the proposed single arm multicenter phase-II trial it is intended to investigate the feasi-bility of adding Avelumab to FOLFIRI plus Cetuximab after 4 cycles (2 months) of treatment with FOLFIRI plus Cetuximab. After 4 more cycles of FOLFIRI plus Cetuximab plus Avelumab the treatment will be de-escalated to Avelumab as a maintenance concept until progression of the disease according to RECIST 1.1 has occurred.

DETAILED DESCRIPTION:
After 4-6 months of doublet chemotherapy a de-escalation to a less toxic regimen is needed for most of the patient with mCRC. The addition of Avelumab to a cytotoxic chemotherapy regimen with FOLFIRI plus cetuximab followed by Avelumab maintenance has not been in-vestigated so far. It is known that FOLFIRI plus cetuximab leads to necrosis and therefore tumor antigens that usually are not presented to the host immune system become recogniza-ble. This effect of a triggered immune system after induction treatment with chemotherapy is currently investigated in other trials. The ongoing IMPALA trial is testing the toll-like receptor (TLR)-9 agonist MGN1703 as maintenance treatment in patients that have responded to an induction doublet chemothera-py. This effect may be enhanced by the fact that Cetuximab in Combination with 5-FU and Irinotecan triggers immunogenic cell death.

The lately published data from the interim analysis of the PACIFIC trial using the anti-PD L1 antibody durvalumab after chemoradiation in stage II non-small cell lung cancer (NSCLC) proofed the concept of an anti-PD L1 antibody as a maintenance treatment after chemoradi-ation. Durvalumab prolonged PFS significantly (HR 0.52, p<0.001).

The study is not limited to MSI-h and should be able to demonstrate Avelumab efficacy in MSS tumors. The lately presented data on the use of atezolizumab plus cobimetinib (NCT01988896) in in heavily pretreated MSS mCRC patients showed a 12-month OS rate of 43% which was higher than the 24% seen for Regorafenib in the pivotal CORECT trial. Therefore it is worthwhile to test this concept in MSS mCRC.

Furthermore part of the cetuximab effect can be attributed to ADCC (antibody derived cellu-lar cyctotoxicity) with again leads to necrosis of tumor cells and the release of antigens. Both effects together may be able to present enough tumor-neo-antigens. To boost the effect, Avelumab is able to inhibit the PD-1 derived inhibition of cytolysis and other tumor cells within the body may be attacked by the immune system which leads to an anti-tumor effect repre-sented by a prolonged PFS and finally OS of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, UICC stage IV adenocarcinoma of the colon or rectum with metastases (metastatic colorectal cancer), metastases primarily non-resectable or surgery refused by the patient
* RAS wild-type tumour status (KRAS and NRAS exon 2, 3, 4) (proven in the primary tumour or metastasis)
* Age ≥18
* ECOG performance status 0-1
* Patients suitable for chemotherapy administration
* Patient's written declaration of consent obtained
* Estimated life expectancy > 3 months
* Presence of at least one measurable reference lesion according to the RECIST 1.1 criteria
* Primary tumour tissue available and patient consents to storage and molecular and genetic profiling of tumour material. Molecular profiling of blood samples is optionally performed.
* Females of childbearing potential (FCBPs) and men must agree to use highly effec-tive contraceptive measures (Pearl index <1) or practice true abstinence from any heterosexual intercourse (true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject) for the duration of the study treatment and for at least 6 months after last administration of study medication. A woman will be considered as being of childbearing potential unless she is at least 50 years old and moreover has gone through menopause for at least 2 years or has been surgically sterilised.
* Adequate bone marrow function:

  * Leukocytes ≥ 3.0 x 109/L with neutrophils ≥ 1.5 x 109/L
  * Thrombocytes ≥ 100 x 109/L
  * Haemoglobin ≥ 5.6 mmol/L (equivalent to 9 g/dL)
* Adequate hepatic function:

  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * ALAT and ASAT ≤ 2.5 x ULN (in the presence of hepatic metastases, ALAT and ASAT ≤ 5 x ULN)
  * INR < 1.5 and aPTT < 1.5 x ULN (patients without anticoagulation). Therapeu-tic anticoagulation is allowed if INR and aPTT have remained stable within the therapeutic range for at least 2 weeks.
  * Adequate renal function:
  * Creatinine clearance (calculated according to Cockcroft and Gault) ≥ 50 mL/min
* Adequate cardiac function: ECG and echocardiogram with a LVEF of ≥ 55%
* No previous chemotherapy for metastatic disease. Patient with need of immediate treatment (high tumour load, symptoms) may have received one application of FOLFIRI prior to study entry.
* Time interval since last administration of any previous neoadjuvant/adjuvant chemo-therapy or radiochemotherapy of the primary tumour in curative treatment intention ≥ 6 months.
* Any relevant toxicities of prior treatments must have resolved

Exclusion Criteria:

* Proof of a RAS mutation (KRAS or NRAS, exons 2, 3, 4 in the tumor (proven in the primary tumor or metastasis) or absence of testing for RAS mutation
* Primarily resectable metastases and the patient wishes for resection
* ≥ Grade II heart failure (NYHA classification)
* Myocardial infarction, balloon angioplasty (PTCA) with or without stenting, and cere-bral vascular accident/stroke within the past 12 months before start of study treat-ment, unstable angina pectoris, serious cardiac arrhythmia according to investigator's judgement requiring medication.
* Pre-existing pulmonary fibrosis or immune pneumonitis
* Active autoimmune disease that might be negatively affected by an immune check-point inhibitor. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation, including allogeneic stem cell transplantation
* Current use of immunosuppressive medication, except for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan pre-medication).
* Pregnancy (absence of pregnancy to be ascertained by a negative beta hCG test) or breast feeding
* Medical or psychological impairments associated with restricted ability to give con-sent or not allowing conduct of the study
* Additional cancer treatment (chemotherapy, radiation, immunotherapy or hormone treatment) during the study treatment in first-line and third-line treatment (treatments that are conducted as part of an anthroposophic or homeopathic treatment approach, e.g. mistletoe therapy do not represent an exclusion criterion)
* Previous chemotherapy for the colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before entering the study
* Toxicity > Grade 1 that has not yet resolved, attributed to a previous treatment or measure for treatment of the mCRC. However, alopecia (all grades) and oxaliplatin-induced neurotoxicity ≤ Grade 2 are acceptable.
* Participation in a clinical study or experimental drug treatment within 30 days prior to study inclusion or within a period of 5 half-lives of the substances administered in a clinical study or during an experimental drug treatment prior to inclusion in the study, depending on which period is longest or simultaneous participation in another study while taking part in the study
* Known hypersensitivity or allergic reaction to any of the following substances: 5-fluorouracil, folinic acid, capecitabine, cetuximab, irinotecan, bevacizumab, avelumab and chemically related substances and/or hypersensitivity to any of the components in the formulations of the aforementioned substances, including known hypersensitivi-ty reactions to monoclonal antibodies NCI CTCAE Grade ≥ 3.
* Known hypersensitivity to Chinese hamster ovary cell (CHO) - cellular products or other recombinant human or humanised monoclonal antibodies
* Patients with known brain metastases. In case of clinical suspicion of brain metastasis a cranial CT or MRI must be performed to rule out brain metastasis before study in-clusion.
* History of acute or subacute intestinal occlusion, inflammatory bowel disease, im-mune colitis or chronic diarrhoea
* Symptomatic peritoneal carcinosis
* Severe, non-healing wounds, ulcers or bone fractures
* Patients with active infection requiring systemic therapy
* Known history of testing positive for HIV or known acquired immunodeficiency syn-drome.
* Active or chronic Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive; sero-logic tests required).
* Requirement for immunisation with live vaccine under the study treatment.
* Haemorrhagic diathesis or known thrombophilia
* Known DPD deficiency (specific screening not required)
* Known glucuronidation deficiency (Gilbert's syndrome) (specific screening not re-quired)
* History of a second primary malignancy during the past 5 years before inclusion in the study or during participation in the study, with the exception of a basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ, if these were treated curatively.
* Known history of alcohol or drug abuse
* Any other severe acute or chronic concomitant disease or medical condition including psychiatric conditions (including recent i.e. within the past year or active suicidal idea-tion or behavior) or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the in-terpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Absent or restricted legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 8 months
  The primary clinical objective is to determine the efficacy of a standard 1st-line regimen (FOLFIRI plus cetuximab) in patients with RAS wild-type mCRC with Avelumab mainte-nance in terms of progression free survival rate after 8 months (according to RECIST 1.1).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 36 months
  Determine safety and tolerability, according to NCI CTC AE v4.03 and to the obtained data on vital signs, clinical parameters (oxygen saturation) and feasibility of the regimen.
Efficacy of experimental Regimen according to response rate | up to 36 months
  Determine the efficacy of the experimental regimen in terms of objective response rate (acc. to RECIST v1.1 and irRE-CIST)
Efficacy of experimental Regimen according to Overall survial | up to 36 months
  Determine the efficacy of the experimental regimen in terms of overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Modest, PD Dr., Study Chair — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig Maximilians University, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided